CLINICAL TRIAL: NCT06172595
Title: 18F-FET (O-(2-[18F]Fluoroethyl)-L-tyrosine) PET in Differentiating Tumour Progression From Pseudoprogression in High Grade Gliomas
Brief Title: FET PET in Differentiating Tumour Progression From Pseudoprogression in High Grade Glioma
Acronym: FET PET in HGG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other); National Neuroscience Institute Singapore (Unknown); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202112-00050
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FET PET (Experimental): Upon recruitment, a single study visit will be scheduled where subjects undergo a limited 18F-FET PET/CT of the brain in SGH.
  After the study visit, from time of recruitment, they will continue their regular clinic visits as clinically indicated, where they will be monitored for at least a year for stability or deterioration. If clinically indicated, they may undergo conventional MRI, alternative MRI imaging and/or histopathological correlation in their respective primary institutions.
  During these follow-up visits, any adverse effects possibly attributed to the 18F-FET PET/CT can also be flagged up.
  Any alternative MRI imaging performed (as part of clinical practice in the respective primary institutions) within 4 weeks of the 18F-FET PET/CT study will also be included in the comparative analysis.
  Interventions: Diagnostic Test: FET PET

INTERVENTIONS:
Diagnostic Test: FET PET — There is only one study visit during which study subjects will undergo a 18F-FET PET/CT in SGH. Following that, they will be followed up as per their routine clinical care. Data collection timepoints will be at 30 days, 4 months, 8 months and 1 year.

SUMMARY:
The goal of this clinical trial is to evaluate the performance characteristics of O-(2-[18F]fluoroethyl)-L-tyrosine (FET) PET in differentiating pseudoprogression from tumour progression in patients with equivocal conventional imaging and determine the sensitivity and specificity of [18F]FET-PET in delineating disease. The main question[s] it aims to answer are:

* whether 18F-FET-PET will demonstrate high diagnostic accuracy to detect true tumour progression
* whether we can optimise the threshold cut-offs for TBRmax and other relevant parameters in discriminating pseudoprogression and disease progression Participants will undergo a limited 18F-FET PET/CT of the brain in SGH.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women, aged 21 years or older at time of screening
* Histologically confirmed diagnosis of malignant glioma (defined as WHO grade III or IV) with previous RT to tumour
* With enlarging contrast-enhancing and/or T2W/FLAIR-hyperintense lesion(s) on MRI within the previous RT field
* Gliomas with Isocitrate dehydrogenase (IDH) wild-type status, as defined on immunohistochemistry
* Subject must consent to undergo all study procedures

Exclusion Criteria:

* Low-grade gliomas (histology grade 1 or 2 by WHO classification)16,17
* Previous bevacizumab or other vascular endothelial growth factor (VEGF) targeting agents or anti-angiogenic treatments.
* Proven cerebral metastases
* IDH-mutated gliomas
* Pregnancy/ breast-feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics of FET PET in differentiating pseudoprogression from tumour progression in patients with equivocal conventional imaging | 1 year
  Sensitivity and specificity of [18F]FET-PET in delineating disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided